CLINICAL TRIAL: NCT00555685
Title: Hypertonic Saline Solution in Decompensated Heart Failure
Brief Title: Hypertonic Saline Solution in Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Edimar Alcides Bocchi, Heart Failure Team Director, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FAPESP 2007/04048-7
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Heart Failure; Renal Failure; Hyponatremia
Keywords: Heart Failure; Renal failure; Hyponatremia
MeSH Terms: conditions — Heart Failure; Renal Insufficiency; Hyponatremia | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Group of patients that will receive hypertonic saline solution (NaCl 7,5%)
  Interventions: Drug: NaCl 7,5% (Hypertonic Saline Solution)
- B (Placebo Comparator): Group of patients that will receive placebo
  Interventions: Drug: NaCl 0,9%

INTERVENTIONS:
Drug: NaCl 7,5% (Hypertonic Saline Solution) — Patients in the intervention arm will receive 100ml of NaCl 7,5, twice daily during 3 days
  Arms: A
Drug: NaCl 0,9% — Patients in the placebo arm will receive 100ml of NaCl 0,9% twice daily during 3 days
  Arms: B

SUMMARY:
Patients with decompensated heart failure have high rates of mortality and morbidity despite recent improvements in diagnosis and treatment. Some aspects of their presentation such as renal failure, hyponatremia and congestive phenomena have received special attention, as they are associated with worse prognosis. The infusion of hypertonic saline solution has been tested in different conditions of cardiovascular collapse. Current evidence indicates that the infusion of hypertonic solution in heart failure patients can provide clinical and haemodynamic improvement. The investigators are testing the hypothesis that the infusion of hypertonic solution in association with diuretics may prevent the occurrence of renal dysfunction in patients with decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Heart failure according to Framingham criteria
* Episode of acute decompensation,with need of in-hospital treatment
* Presence of congestive phenomena

Exclusion Criteria:

* Patient denial
* Left-ventricle ejection fraction over 0,4, as measure by transthoracic echocardiography
* Rheumatic disease
* Restrictive cardiomyopathy
* Alcohol abuse
* Chronic obstructive pulmonary disease
* Cancer
* Pulmonary embolism during the last 6 months
* Surgical procedures or acute illness during the last 30 days
* Chronic or acute infection
* Any other circumstance that may hamper patient prognosis for the next 6 months
* Serum creatine over 3.0mg/dL
* Serum potassium over 5.5 mEqs/L
* Any specific condition associated to the acute episode of decompensation, such as new onset cardiac arrhythmias, heart ischemia, infection, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of renal disfunction | During hospital admission

SECONDARY OUTCOMES:
Improvement of hyponatremia | During hospital admission
Improvement of congestive phenomena | During hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Edimar A Bocchi, Professor, Principal Investigator — Heart Failure (InCor) University of São Paulo Medical School
Locations (1):
- Heart Institute of São Paulo University Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Rocha-e-Silva M, Poli de Figueiredo LF. Small volume hypertonic resuscitation of circulatory shock. Clinics (Sao Paulo). 2005 Apr;60(2):159-72. doi: 10.1590/s1807-59322005000200013. Epub 2005 Apr 26. PMID 15880253
- [Background] Licata G, Di Pasquale P, Parrinello G, Cardinale A, Scandurra A, Follone G, Argano C, Tuttolomondo A, Paterna S. Effects of high-dose furosemide and small-volume hypertonic saline solution infusion in comparison with a high dose of furosemide as bolus in refractory congestive heart failure: long-term effects. Am Heart J. 2003 Mar;145(3):459-66. doi: 10.1067/mhj.2003.166. PMID 12660669
- [Result] Issa VS, Bacal F, Mangini S, Carneiro RM, Azevedo CH, Chizzola PR, Ferreira SM, Bocchi EA. Hypertonic saline solution for renal failure prevention in patients with decompensated heart failure. Arq Bras Cardiol. 2007 Oct;89(4):251-5. doi: 10.1590/s0066-782x2007001600007. English, Portuguese. PMID 17992382
- [Derived] Issa VS, Andrade L, Ayub-Ferreira SM, Bacal F, de Braganca AC, Guimaraes GV, Marcondes-Braga FG, Cruz FD, Chizzola PR, Conceicao-Souza GE, Velasco IT, Bocchi EA. Hypertonic saline solution for prevention of renal dysfunction in patients with decompensated heart failure. Int J Cardiol. 2013 Jul 15;167(1):34-40. doi: 10.1016/j.ijcard.2011.11.087. Epub 2012 Jan 12. PMID 22243938